CLINICAL TRIAL: NCT00935857
Title: Balloon Colonoscopy Versus Repeat Standard Colonoscopy for Prior Incomplete Colonoscopy: A Randomized Controlled Trial
Brief Title: Balloon Colonoscopy for Incomplete Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significant difference at interim analysis
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rajesh Keswani, Assistant Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00008540
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Diverticulosis
Keywords: Balloon Enteroscopy; Looping
MeSH Terms: conditions — Diverticulum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon Colonoscopy (Experimental): Colonoscopy using the single balloon colonoscopy system (novel endoscope to facilitate difficult colonoscopy).
  Interventions: Device: Single Balloon Colonoscopy
- Standard Colonoscopy (Active Comparator): Colonoscopy using a standard adult colonoscope
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: Single Balloon Colonoscopy — Use of the single balloon enteroscopy system (enteroscope and balloon-overtube) to complete colonoscopy.
  Arms: Balloon Colonoscopy
Device: Standard Colonoscopy — Use of the standard adult colonoscope to complete colonoscopy.
  Arms: Standard Colonoscopy

SUMMARY:
Patients with a prior incomplete colonoscopy will be enrolled in this study. Patients will be randomized to either an initial repeat attempt with a standard colonoscope or the single balloon enteroscope. If the procedures is unsuccessful, the patient can be crossed-over to the other group. The primary endpoint of the study is a complete colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is a well-established practice utilized for the evaluation of lower gastrointestinal tract diseases including, mostly commonly, the screening for colorectal polyps and cancer. Despite improvements in endoscope technology, a significant minority of procedures (up to 10%) can not be safely completed due to a variety of patient factors and technical difficulties. These factors primarily include prior abdominal surgeries resulting in adhesions, severe diverticular disease, inadequate bowel cleansing, and patient discomfort.

Options for an incomplete colonoscopy include several endoscopic and non-endoscopic modalities. Non-endoscopic modalities include radiologic studies such as CT/MRI colonography as well as a retrograde barium study. Relative disadvantages of these modalities is the inability to remove colonic polyps, perform biopsies, and in the case of barium studies, a lower sensitivity for pathology. Alternative endoscopic modalities have been described that may assist in successfully completing colonoscopy Of these alternative methods, balloon-overtube assisted colonoscopy is the most promising, but this method has not been studied in a randomized, controlled fashion. In this study, we aim to compare balloon-overtube assisted colonoscopy versus standard colonoscopy for patients with prior incomplete colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* prior colonoscopy that was incomplete within the previous 12 months or their two most recent colonoscopies (performed at any time interval) were incomplete

Exclusion Criteria:

* incomplete colonoscopy due only to poor bowel preparation or inadequate sedation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh N Keswani, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment completed.
Pre-assignment Details: Early termination at 30 patients due to clinically significant differences at midpoint of study.
  Patients in the Standard Colonoscopy group could cross-over to the Balloon Colonoscopy group after 20 minutes of procedure time but they were not included in further analysis after cross-over.
Groups:
- Balloon Colonoscopy: Colonoscopy using the single balloon enteroscope system.
Period: Overall Study
Arm/Group | Balloon Colonoscopy | Standard Colonoscopy
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: An interim analysis was performed at 30 patients as described in initial protocol. The study was terminated at the interim analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Colonoscopy | Standard Colonoscopy | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.5) | 59.9 (10.0) | 59.2 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Complete Colonoscopy to the Cecum
Description: Number of patients with a complete colonoscopy to the cecum
Time Frame: Day of Procedure
Population: Per Protocol, Terminated at Interim Analysis
Measure: Number; unit: patients
Arm/Group | Balloon Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 14 | 16
patients | 13 | 8

2. Secondary Outcome: Time (Minutes) to Cecum
Description: Time, in minutes, until reaching cecum in each arm.
Time Frame: Day of Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Balloon Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 14 | 16
minutes | 24 (15) | 22 (18)

3. Secondary Outcome: Procedural Complications
Description: Number of patients with any procedural complications as assessed 7 days after procedure.
Time Frame: 7 days post procedure
Measure: Number; unit: participants
Arm/Group | Balloon Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 14 | 16
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week after completion of endoscopy procedure.
Description: All subjects were called 1 week after completion of procedure to assess for adverse events.
Groups:
- Standard Colonoscopy: Patients who are randomized to received standard colonoscopy as initial treatment.
- Single Balloon Colonoscopy: Patients who are randomized to received single balloon colonoscopy as initial treatment.
Arm/Group | Standard Colonoscopy | Single Balloon Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
Early termination due to interim analysis showing statistical difference; single operator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes